CLINICAL TRIAL: NCT02153723
Title: Pharmacological Treatment of Rett Syndrome With Glatiramer Acetate (Copaxone)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Rett Syndrome Research Trust (Other)
Responsible Party: Principal Investigator, Aleksandra Djukic, Associate Professor of Clinical Neurology and Clinical Pediatrics, Director, Tri State Rett Syndrome Center, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-05-117
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Rett Syndrome
Keywords: Treatment trial, Rett syndrome, Glatiramer acetate
MeSH Terms: conditions — Rett Syndrome | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Copaxone (Experimental): Dose escalation:
  Study drug will be administered once a week for 4 weeks, twice a week for 4 weeks and daily for 24 weeks. Drug is administered as a subcutaneous injection.
  Interventions: Drug: Glatiramer Acetate

INTERVENTIONS:
Drug: Glatiramer Acetate
  Other Names: Copaxone

SUMMARY:
A phase 2 open label trial to test a potential drug treatment for Rett syndrome, the leading known genetic cause of severe neurological impairment in girls. The drug, Copaxone (generic name - Glatiramer acetate) is medication FDA approved for the treatment of multiple sclerosis. Copaxone's high safety profile has been documented in large cohorts of patients for more than 12 years.

DETAILED DESCRIPTION:
Background/rationale for the study:

In Rett syndrome brain cells aren't actually lost, instead poor maturation of connections between brain cells (synapses) prevents effective neurological functioning, and is the main morphological feature of the disease. The MeCP2 gene plays a major role in transcriptional regulation of other genes, one of which is the gene encoding brain-derived neurotrophic factor (BDNF).

The disease progression and severity of symptoms is directly affected by the level of BDNF expression. An increase of BDNF levels (by genetic manipulations or pharmacological agents) leads to delayed onset of Rett syndrome-like symptoms in experimental models; rescued gait/mobility, improved quality of life and increased survival rates.

Copaxone treatment by subcutaneous injection caused elevation of BDNF levels. Quantitative immunofluorescence assays showed about a twofold increase in neuronal expression of BDNF following Copaxone treatment.

We expect that an increase in BDNF levels with Copaxone administration will stimulate communication between brain cells (synaptic maturation), which will lead to amelioration of symptoms (motor functions/gait, cognitive functions, breathing, encephalopathy and improve quality of life) for girls with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with genetically confirmed Rett Syndrome (RTT)
* Age: 10 or more years old. Selection of the age is based on the available evidence of the safety of Glatiramer Acetate (GA) in this group, and the relative homogeneity/stability of the phenotype, which is not expected to spontaneously change within a 6 month period at this age
* Ambulatory (with our without support)

Exclusion Criteria:

* Prolonged Qtc (obtained within 30 days prior to enrollment)
* Presence of co morbid non-Rett related disease
* Presence of immunodeficiency requiring intravenous immunoglobulin 3 (IVIG 3) months prior to enrollment
* Allergy/sensitivity to GA or mannitol
* Inability or unwillingness of legal guardians to give written informed consent

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Djukic A, Holtzer R, Shinnar S, Muzumdar H, Rose SA, Mowrey W, Galanopoulou AS, Shinnar R, Jankowski JJ, Feldman JF, Pillai S, Moshe SL. Pharmacologic Treatment of Rett Syndrome With Glatiramer Acetate. Pediatr Neurol. 2016 Aug;61:51-7. doi: 10.1016/j.pediatrneurol.2016.05.010. Epub 2016 May 27. PMID 27363291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited between Aug 2014-Jan 2015, from the population treated at the Rett Center at Montefiore.
  Of 11 screened subjects, 10 met the inclusion/exclusion criteria and completed the trial. One patient was excluded due to prolonged QTc.
  Data analysis was performed after the first 10 participants completed the study.
Groups:
- Copaxone: Dose escalation:
  Study drug will be administered once a week for 4 weeks, twice a week for 4 weeks and daily for 24 weeks. Drug is administered as a subcutaneous injection.
  Glatiramer Acetate
Period: Overall Study
Arm/Group | Copaxone
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants were female, ambulatory, and had been previously diagnosed with Rett syndrome.
Arm/Group | Copaxone
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were female
  Participants
    Female | 10
    Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity as Measured by GAITRite System
Description: To perform quantitative gait assessments a computerized walkway (457 × 90.2 × 0.64cm) with embedded pressure sensors (GAIT Rite system) was used. Subjects walked on the walkway for two trials, while wearing comfortable footwear.
Time Frame: Baseline and Final week of treatment (week 32)
Population: All 10 patients were females with genetically confirmed Rett syndrome. All were at least 10 years old and ambulatory (walking without assistance at the time of their enrollment).
Measure: Median (Inter-Quartile Range); unit: cm/sec
Arm/Group | Copaxone
Number analyzed (Participants) | 10
cm/sec
  Baseline | 62.7 [42.3 to 103.2]
  Final week of treatment (week 32) | 84.3 [58.1 to 119.3]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.03, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 21.6

2. Secondary Outcome: Breath Hold Index (Number of Breath Holds Per Hour; Assessed in the Sleep Monitoring Lab)
Description: Breath hold index is defined as number of breath holds/hour. Respirations were monitored with sleep monitoring equipment during the daytime at the polysomnography laboratory with additional oronasal airflow, electromyography (EMG), EEG and video monitoring to confirm wakefulness during the period of study.
Time Frame: Baseline and during final week of treatment (week 32)
Population: One of the 10 enrolled patients experienced panic attack during the respiratory function testing so that session was discontinued. This left 9 participants for final analysis.
Measure: Median (Inter-Quartile Range); unit: number of breath holds/hour
Arm/Group | Copaxone
Number analyzed (Participants) | 9
number of breath holds/hour
  Baseline | 3.8 [2.3 to 7.3]
  Final week of treatment (week 32) | 1.6 [0.3 to 2.0]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.03, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.0

3. Secondary Outcome: Breath Hold Time (Assessed in the Sleep Monitoring Lab)
Description: Breath Hold Time is defined as percentage of time spent holding the breath in a specific time unit. It is measured by a standard medical technique where belts are placed on the chest and abdomen to record movement and sensors are used to record nasal flow. Wake respiration was monitored with sleep monitoring equipment during the daytime at the polysomnography laboratory with additional oronasal airflow, EMG, EEG and video monitoring to confirm wakefulness during the period of study.
Time Frame: Baseline and Final week of treatment (week 32)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Copaxone
Number analyzed (Participants) | 9
percentage of time
  Baseline | 1.8 [0.8 to 2.3]
  Final week of treatment (week 32) | 0.4 [0.1 to 0.8]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.1

4. Secondary Outcome: Visual Memory Novelty Score as Assessed by TX300 Tobii Computer.
Description: Eye-tracking is considered an indication of visual memory. Eye-tracking data was recorded at 300 Hz sampling rate using a Tobii T300 computer (Tobii Technology, Danderyd, Sweden). The actual data given by the computer represents the percentage of time spent looking at a novel visual target - this is called the novelty score. Visual memory, as indexed by the novelty score, is the percentage of time spent looking at a novel target during the test ("visual paired comparison paradigm"). Duration of testing was 2 minutes.
Time Frame: Baseline and Final week of treatment (week 32)
Population: Only 7 of the 10 recruited participants were able to complete the cognitive assessment. The remaining 3 participants could not be tested due to technical reasons.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Copaxone
Number analyzed (Participants) | 7
percentage of time
  Baseline | 42.4 [39.5 to 61.0]
  Final week of treatment (week 32) | 62.4 [55.7 to 65.8]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.08, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 15.9

5. Secondary Outcome: Visual Attention (Number of Fixations) Assessed by Eye-tracking TX300 Tobii Computer.
Description: Visual attention is indexed by duration and number of fixations on novel target on testing. The standard method of assessing visual attention in neuropsychology is by measuring:
  A)number of fixations (how many times the subject looks at each of the 2 visual targets). The higher number of fixations, the more attentive the subject to that visual target.
  B) duration of fixations in seconds (the longer the fixation the more attentive). Duration of fixations correlates with intelligence: the smarter the person is the shorter his fixations are.
  Eye-tracking data was recorded at 300 Hz sampling rate using a Tobii T300 (Tobii Technology AB, Danderyd, Sweden). The measured index is called the Novelty Score which indicates the percentage of time spent looking at novel visual target. Duration of testing session was 2 minutes.
Time Frame: Baseline and Final week of treatment (week 32)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: number of fixations
Arm/Group | Copaxone
Number analyzed (Participants) | 7
number of fixations
  Baseline | 19.4 [8.0 to 20.8]
  Final week of treatment (week 32) | 16.2 [11.0 to 27.4]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.86, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.8

6. Secondary Outcome: Visual Attention (Fixation Length) Assessed by Eye-tracking TX300 Tobii Computer.
Description: The standard method of assessing visual attention in neuropsychology is by measuring:
  A)number of fixations (how many times the subject looks at each of the 2 visual targets). The higher number of fixations, the more attentive the subject to that visual target.
  B) duration of fixations in seconds (the longer the fixation the more attentive). Duration of fixations correlates with intelligence: the smarter the person is the shorter his fixations are.
  Eye-tracking data was recorded at 300 Hz sampling rate using a Tobii T300 (Tobii Technology AB, Danderyd, Sweden). The measured index is called the Novelty Score which indicates the percentage of time spent looking at novel visual target. Visual attention is indexed by number of fixations on novel target on test.
  Duration of testing session was 2 minutes.
Time Frame: Baseline and Final week of treatment (week 32)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Copaxone
Number analyzed (Participants) | 7
seconds
  Baseline | 0.46 [0.26 to 0.64]
  Final week of treatment (week 32) | 0.35 [0.18 to 0.46]
Statistical Analysis 1: Comparison: Copaxone; Test type: Other — Wilcoxon signed rank sum test; p = 0.44, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00

ADVERSE EVENTS:
Arm/Group | Copaxone
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copaxone (N=10)
laboratory result (elevated CPK) without clinical correlate, transitory (Musculoskeletal and connective tissue disorders) | 1 (1) — not sympromatic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No